CLINICAL TRIAL: NCT05209581
Title: Assessment of Visual Acuity of the Refugee Population
Brief Title: Assessment of Visual Acuity in Refugee Population
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: DUTh REC/4/16-12-2021
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Visual Acuity; Refractive Errors; Low Vision; Vision Disorders
Keywords: distance visual acuity; refugee; immigrant
MeSH Terms: conditions — Refractive Errors; Vision, Low; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Adult refugees/immigrants living in accommodation structures
  Interventions: Diagnostic Test: Distance Visual Acuity Examination

INTERVENTIONS:
Diagnostic Test: Distance Visual Acuity Examination — Best spectacle-corrected distance visual acuity of refugees/immigrants will be examined via a web-based digital visual acuity chart

SUMMARY:
The present research process is a prospective clinical study that will be conducted under the auspices of the Democritus University of Thrace (DUTH) in the open accommodation structure for refugees and immigrants of Kavala, Kavala, Greece, and the Pre-Removal Detention Center (PROKEKA) for Foreigners of Kos, Kos, Greece. The study aims to assess the basic ophthalmological condition of the refugee/immigrant population and is developed in two main areas:

1. The recording of the ophthalmological care that the refugee/immigrant has received until his/her inclusion in the study through a structured questionnaire (eg previous examinations, spectacle utilization, pharmaceutical or other interventions, etc.)
2. The measurement of monocular best-spectacle corrected visual acuity in both eyes using a web-based visual acuity chart.

Adult participants living in the two aforementioned centers will be recruited in a consecutive-if-eligible basis. All age groups will be proportionally represented (proportional age distribution).

DETAILED DESCRIPTION:
Study protocol will adheres to the tenets of the Helsinki Declaration and written informed consent translated in the language of each examinee will be obtained by all participants. Subsequently, participants will complete a questionnaire about demographic and general clinical information.

Then, the best spectacle-corrected distance visual acuity of each participant's both eyes will be evaluated monocularly via a web-based digital chart in a high-resolution screen. The same environmental lighting conditions and the same screen brightness will be applied. The examination will be performed at the same predetermined viewing distance.

Finally, according to each participant's visual acuity, appropriate instructions will be given for the improvement of his/her eye care.

ELIGIBILITY:
Inclusion Criteria:

* Adult refugees or immigrants

Exclusion Criteria:

* Visual acuity lower than 1.0 LogMAR
* Age <18 years
* Refugees or immigrants living in the accommodation structures without yet having the appropriate legal documents

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal- and low-vision adult refugees or immigrants living in accommodation structures
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Best spectacle-corrected distance visual acuity | 1 week
  Best spectacle-corrected distance visual acuity of refugees will be examined via a web-based digital visual acuity chart

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Democritus University of Thrace
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: Undecided